CLINICAL TRIAL: NCT04170114
Title: Comparison of the Efficacy of Comprehensive Respiratory Physiotherapy in Children With Cystic Fibrosis and Non-Cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bvuhucgun02
Record Dates: First submitted 2019-11-12; First posted 2019-11-20 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Cystic Fibrosis; Bronchiectasis
Keywords: Cystic Fibrosis; Bronchiectasis; Respiratory Physiotherapy; Pulmonary Function; Exercise Capacity; Six Minute Walk Test; Muscle Strength
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cystic Fibrosis (Experimental): Children with cystic fibrosis
  Interventions: Other: Comprehensive Respiratory Physiotherapy
- Bronchiectasis (Experimental): Children with bronchiectasis
  Interventions: Other: Comprehensive Respiratory Physiotherapy

INTERVENTIONS:
Other: Comprehensive Respiratory Physiotherapy — All patients will receive comprehensive respiratory physiotherapy training by the physiotherapist. All patients will undergo comprehensive respiratory physiotherapy techniques twice daily for 8 weeks.
  Comprehensive respiratory physiotherapy programme will include diaphragmatic breathing exercise, thoracic expansion exercises, incentive spirometer exercise (Triflo), oscillatory PEP (Flutter), postural drainage, coughing techniques and teaching respiratory control.

SUMMARY:
The effect of comprehensive respiratory physiotherapy applications on respiratory function, functional capacity and peripheral muscle strength in children with cystic fibrosis and non-cystic fibrosis will be compared.

DETAILED DESCRIPTION:
Bronchiectasis may be a congenital cause such as cystic fibrosis (CF) or non-cystic fibrosis such as primary ciliary dyskinesia, post-infectious conditions, aspiration and immunodeficiency; It is a disease characterized by irreversible dilatation of airways. Symptoms; purulent sputum production, chronic cough, hemoptysis, recurrent fever and pleurisy. Mucociliary clearance disorder secondary to inflammation and involvement of exocrine glands in CF plays a major role in the development of symptoms; In non-cystic fibrosis bronchiectasis (NCFB), the development of similar symptoms may occur regardless of these reasons. However, in the examinations of CF, proximal airways; In NCFB, distal airways have been affected more intensively. As part of pulmonary rehabilitation, comprehensive respiratory physiotherapy (CRP) has an important role in the treatment and management of bronchiectasis. Airway cleaning techniques, approaches to reducing respiratory work, and patient education form the basis of CRP and play an active role in the treatment and management of the disease. In the literature, there are studies in which the effects of CRP are given in both CF and NCFB patients and studies comparing evaluation results in both groups without treatment. However, no study was found to compare the efficacy of CRP in these two groups of diseases. Therefore, in this study, the investigators aimed to investigate the differences between the efficacy of CRP among the groups in children with CF and NCFB.

ELIGIBILITY:
Inclusion Criteria:

* Being between 6-18 years old
* Clinically diagnosed as cystic fibrosis or non-cystic fibrosis bronchiectasis

Exclusion Criteria:

* Previous history of lung or liver transplantation
* Have had an acute exacerbation in the last month and / or have a history of hospitalization
* Having a diagnosis of orthopedic problems affecting mobility or a history of musculoskelatal surgery

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | 8 Weeks
  FVC will be measured using basic spirometry and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
Forced Expiratory Volume in 1 second (FEV1) | 8 Weeks
  FEV1 will be measured using basic spirometry and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
Peak Expiratory Flow (PEF) | 8 Weeks
  PEF will be measured using basic spirometry and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
Respiratory Muscle Strength - MIP | 8 Weeks
  Maximum Inspiratory Pressure (MIP) will be measured using MicroRPM portable manometer and the unit will be expressed in mmHg
Respiratory Muscle Strength - MEP | 8 Weeks
  Maximum Expiratory Pressure (MEP) will be measured using MicroRPM portable manometer and the unit will be expressed in mmHg
Six-minute walk test distance | 8 Weeks
  Distance walked in six minutes will be recorded in meters. Test will be conducted according to the guideline of American Thoracic Society (ATS)
M. Quadriceps strength | 8 Weeks
  sometric M. Quadriceps strength (kg) will be measured using electronic hand held dynamometer in sitting position.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif Universitesi, Department of Physiotherapy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided